CLINICAL TRIAL: NCT04923737
Title: Immunomodulatory Effects of Dexmedetomidine Infusion After Laparoscopic Major Abdominal Surgeries: Randomized Controlled Study
Brief Title: Immunomodulatory Effects of Dexmedetomidine Infusion
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Alexandria University (Other)
Responsible Party: Principal Investigator, rehab zayed, Assisstant Professor of Anesthesia, Alexandria University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0304767
Record Dates: First submitted 2021-06-07; First posted 2021-06-11 (Actual); Last update posted 2022-06-01 (Actual); Status verified 2022-05

CONDITIONS: Major Abdominal Surgery
MeSH Terms: interventions — Dexmedetomidine; Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine group (Active Comparator): patients will receive a loading dose of IV Dexmedetomidine1μg/kg slowly just before induction of anesthesia, then Dexmedetomidine infusion started at a rate of 0.5μg/kg/h.
  Interventions: Drug: Dexmedetomidine
- Control group (Placebo Comparator): patients will receive an equal volume of 0.9% sodium chloride (both the loading, and the infusion
  Interventions: Drug: 0.9% sodium chloride

INTERVENTIONS:
Drug: Dexmedetomidine — patients will receive a loading dose of IV Dexmedetomidine1μg/kg slowly just before induction of anesthesia, then Dexmedetomidine infusion started at a rate of 0.5μg/kg/h.
  Arms: Dexmedetomidine group
Drug: 0.9% sodium chloride — patients will receive an equal volume of 0.9% sodium chloride (both the loading, and the infusion
  Arms: Control group

SUMMARY:
Anesthetic management may affect both immunostimulatory and immunosuppressive mechanisms directly by modulating immune cell function or indirectly by attenuating the stress response, Thus, the choice of anesthetic technique may affect clinical outcomes by perturbing the balance between pro- and anti-inflammatory responses,anesthetics favoring this delicate balance are thus desirable as their use may reduce postoperative complications and mortality

ELIGIBILITY:
Inclusion Criteria:

* scheduled for elective laparoscopic major abdominal surgeries;
* ASA class II-III

Exclusion Criteria:

- 1- Patients with severe infection or diseases in respiratory system 2- Patients with severe arrhythmia or bradycardia 3- Patients with severe diseases in liver, kidney, endocrine or immune system. 4- Patients with history of uncontrolled hypertension, A-V conduction block. 5- Patients who had administrated the α-adrenergic agonists or β-receptor antagonist.

6- Patients who received the chemotherapy, radiotherapy, or immunotherapy within one month before operation 7- Patients who had feverbefore operation

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-01-01 (Actual); Primary Completion 2022-05 (Estimated); Study Completion 2022-05 (Estimated)

PRIMARY OUTCOMES:
immune-modulatory effects | three days after surgery
  serum concentrations of C-reactive protein (CRP) level ,The pro-inflammatory cytokines interleukin (IL)-1β, and IL-6 and anti-inflammatory cytokines IL-10 will be measured at four times: T0 (before anesthesia), T1 (1 h after surgery), T2 (24 h after surgery) and T4 (72 h after surgery

CONTACTS AND LOCATIONS:
Overall Officials: rehab A. Abd Elaziz, Ass.Prof., Principal Investigator — Alexandria University
Locations (1):
- Rehab Abd Elraof Abd Elaziz, Alexandria, Egypt